CLINICAL TRIAL: NCT07050836
Title: Contrast Enhanced Ultrasound in Neurosurgery to Improve Glioma Visualization and Border Demarcation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-0399.cc
Record Dates: First submitted 2025-04-30; First posted 2025-07-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Glioma (Any Grade) in the Brain; Glioma
Keywords: brain tumor, resection, glioma
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brain tumor surgery with Definity contrast and Contrast Enhanced Ultrasound (Experimental)
  Interventions: Combination Product: Definity contrast during ultrasound

INTERVENTIONS:
Combination Product: Definity contrast during ultrasound — Definity contrast injection given just prior to brain tumor surgery. Contrast enhanced ultrasound during brain tumor surgical resection to aid in brain tumor visualization.

SUMMARY:
This study plans to learn more about using contrast enhanced ultrasound (CEUS) in brain tumor surgery.

The goal of glioma brain tumor surgery is to remove as much of the glioma as possible. Tumor tissue that is close to normal brain tissue can look very similar. This can make it difficult for the surgeon to remove all the tumor. In this study, we hope to learn if using CEUS during brain tumor surgery will allow the brain surgeon to better see and remove all the tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign and date the consent form
* Stated willingness to comply with all study procedures and be available for the duration of the study
* Be a male or female aged 18-95
* Have a planned standard of care surgery for presumed primary or known recurrent glioma
* WHO performance status </= 2 (equivalent Karnofsky Performance Status, KPS>/= 70)
* Patient of childbearing potential must have a negative pregnancy test within 14 days of inclusion

Exclusion Criteria:

* Patient at high risk of surgical site infection (e.g., 2 or more previous craniotomies/neurosurgery within the last 3 months, poor skin condition, and/or previously infected surgical field, or any other condition that is of increased infectious risk in the opinion of the neurosurgeon)
* Known history of hypersensitivity reactions to perflutren lipid microsphere components or to any of the inactive ingredients in the contrast agent.
* Patient with known or suspected active or chronic infections.
* Patient with known significant cardiac disease, known to have right-to-left shunts, severe pulmonary hypertension (pulmonary artery pressure > 90 mm Hg), uncontrolled systemic hypertension, or adult respiratory distress syndrome.
* Pregnant, or breastfeeding patient.
* Patient with known sickle cell disease.
* Any other serious patient medical or psychological condition that may interfere with adequate and safe delivery of treatment and care.
* Patients under guardianship, curatorship, under legal protection or deprived of liberty by an administrative or judicial decision.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | Up to 3 days
  This study plans to learn more about using contrast enhanced ultrasound (CEUS) to better identify normal brain from tumor in brain tumor surgery.
  The goal of brain tumor surgery is to remove as much of the tumor as possible. Tumor tissue that is close to normal brain tissue can look very similar. This can make it difficult for the surgeon to remove all the tumor. In this study, we hope to learn if using CEUS during brain tumor surgery will allow the brain surgeon to better see and remove all the tumor tissue.
  The ability of CEUS to improve visualization of brain tumor during surgery will be measured by the surgeon during surgery. The surgeon will also take images of the surgery site during surgery with the contrast enhanced ultrasound machine. These images will be studied later to determine if CEUS improves the surgeons ability to better visualize tumor during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: D. Ryan Ormond, MD PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided